CLINICAL TRIAL: NCT00384501
Title: Intacs for the Treatment of Keratoconus
Brief Title: Management of Patients With Keratoconus With Intacs
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of Crete (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PEPAGNI-6175
Record Dates: First submitted 2006-10-05; First posted 2006-10-06 (Estimated); Last update posted 2006-10-06 (Estimated); Status verified 2006-10

CONDITIONS: Keratoconus
Keywords: keratoconus; Intacs
MeSH Terms: conditions — Keratoconus

INTERVENTIONS:
Device: Intacs

SUMMARY:
Purpose To evaluate long-term follow up of Intacs microthin prescription inserts (Addition Technology Inc, Fremont, Calif) for the management of keratoconus.

Design A long-term (five years) retrospective, follow-up study

DETAILED DESCRIPTION:
Subjects and Methods

Ethical committee approval was obtained for the original trial, and patients were asked to sign an informed consent form (in accordance with Institutional guidelines and to the Declaration of Helsinki) before treatment and for further follow-up examinations. The registration information for this clinical trial is available to the public through the National Institute of Health database.

The surgical procedure was done under topical anesthesia. Two Intacs segments of 0.45-mm thickness were inserted so as to embrace the steepest keratoconus meridian, according to the topographic image, aiming at maximal flattening.

The corneal thickness was measured intraoperatively at the incision site and peripherally in the cornea along the ring placement markings with ultrasonic pachymetry (Sonogage, Cleveland, Ohio, USA). Using a diamond knife, set at 70% of the thinnest corneal measurement, a 0.9-mm radial incision was formed, and corneal pockets were created using two Sinskey hooks and a Suarez spreader. Two corneal tunnels were then formed using clockwise and counterclockwise dissectors under suction created by a vacuum-centering guide. The two polymethyl methacrylate (PMMA) segments (0.45-mm thickness) were implanted in the respective corneal tunnels, maintaining a space of approximately 2.0-mm between their ends and 1.5 mm between the opposite edge of each segment and the edge of the incision. The incision site was sutured using a single 10/0 nylon stitch.

Postoperative evaluation Postoperatively, all eyes received antibiotic/steroid combination eye drops 4 times per day for 2 weeks. In addition, all patients were instructed to use preservative-free artificial tears frequently. The sutures were removed 2 weeks after surgery.

Group differences for continuous variables were tested using the paired Student t tests. The change in manifest refraction (spherical equivalent) (MRSE) and topographic k values and topographic astigmatism were plotted over time to determine long-term stability, and the difference as a function of time was analyzed using paired 2-tailed t tests (at time intervals of preoperative to 1 month, 1 to 3 months, 3 to 6 months, 6 to 12 months, and every year of follow up period). Results are presented as means + standard deviation [SD]. A P value less than .05 was regarded as statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* All patients had clear central corneas and contact lens intolerance (rigid gas permeable contact lenses intolerance, frequent contact lens displacement, unsatisfactory visual acuity),

Exclusion Criteria:

* history of herpes keratitis; diagnosed autoimmune disease; and systemic connective tissue disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25
Dates: Start 2000-01; Study Completion 2006-07

PRIMARY OUTCOMES:
refractive stability, UCVA, BSCVA, complications

CONTACTS AND LOCATIONS:
Overall Officials: George D Kymionis, M.D., Ph.D, Principal Investigator — University of Crete

REFERENCES:
- [Result] Alio JL, Shabayek MH, Artola A. Intracorneal ring segments for keratoconus correction: long-term follow-up. J Cataract Refract Surg. 2006 Jun;32(6):978-85. doi: 10.1016/j.jcrs.2006.02.044. PMID 16814056